CLINICAL TRIAL: NCT00574197
Title: Assessment of Gastrointestinal Tolerability and Efficacy of Enteric-coated Mycophenolate Sodium (Myfortic®) in Heart Transplant Recipients
Brief Title: Enteric-coated Mycophenolate Sodium (Myfortic®) in Heart Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Lawrence Czer, MD, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9810
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Gastrointestinal Symptoms; Heart Transplantation
Keywords: Heart Transplant; gastrointestinal; Cellcept; Myfortic; GI; GI symptoms with Mycophenolate Mofetil post heart transplant
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enteric-coated Mycophenolate Sodium (Myfortic) (Other): 1440mg/day (720mg by mouth, twice a day) of enteric-coated Mycophenolate Sodium (Myfortic) for 6 months
  Interventions: Drug: Mycophenolate Sodium

INTERVENTIONS:
Drug: Mycophenolate Sodium — 1440mg/day (720mg by mouth, twice a day)
  Other Names: Myfortic

SUMMARY:
Mycophenolate sodium (Myfortic®) is a newly developed enteric-coated tablet version of mycophenolate mofetil (Cellcept®) which is currently used as therapy for the prevention of transplant rejection. Myfortic® was developed to improve the gastrointestinal tolerability of Cellcept®. The new enteric-coated, Myfortic® is presently FDA approved for the prevention of acute kidney rejection only. There is no clinical data of its use in heart transplant patients.

DETAILED DESCRIPTION:
This is an open-labeled, prospective, non-randomized pilot-phase study of the enteric-coated, Myfortic® versus the non enteric-coated, Cellcept® in patients who are within 5 years of having undergone heart transplant surgery who are currently taking Cellcept®. After the initial screening, 20 patients who fulfill the inclusion criteria and report symptoms of gastrointestinal side-effects while taking Cellcept will be switched to Myfortic. All 20 patients will be followed closely over a period of 6 months following enrollment. Concomitant immunosuppressive therapy will continue in all patients per standard treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex aged 18 and above who have undergone successful orthotopic heart transplant surgery.
2. Patients who are currently taking Cellcept® and experiencing gastrointestinal side-effects from this standard therapy.
3. Individuals on Cellcept® with total dosage of 2 mg a day or less would be eligible to participate.
4. Patients who are able to give written informed consent.

Exclusion Criteria:

1. Patients with an absolute neutrophil count <1500 cells/mm3, and/or leukocytopenia (<2500 cells/mm3), thrombocytopenia (<75,000 cells/mm3) and significant anemia (hemoglobin < 6g/dl) at the time of potential enrollment.
2. Women of childbearing potential not using the contraception method(s), as well as women who are breastfeeding.
3. Known sensitivity to the study drug or class of the study drug.
4. Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study.
5. Use of any other investigational agent in the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernst Schwarz, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars- Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enteric-coated Mycophenolate Sodium (Myfortic)
Started | 11
Completed | 6
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Enteric-coated Mycophenolate Sodium (Myfortic)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: GI Tolerability as Measured by GSRS
Description: Side-effects using the GSRS (Gastrointestinal Symptoms Rating Scale)
  GSRS has 15 items, each rated on a 7-point scale from 1 (no discomfort) to 7 (very severe discomfort). GSRS total minimum value is 15; maximum value is 105. Higher scores represent greater discomfort.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enteric-coated Mycophenolate Sodium (Myfortic)
Number analyzed (Participants) | 6
score on a scale
  GSRS at baseline | 55.67 (15.49)
  GSRS at 6 months | 34.17 (19.47)

2. Secondary Outcome: Number of Biopsy Proven Acute Rejection, Graft Loss and Death Due to Rejection.
Description: Number of biopsy proven acute rejection, graft loss, and death due to rejection.
  Number of rejection episodes where rejection is defined as Grade 1B or higher on myocardial biopsy as measured by the 1990 Grading System of the International Society of Heart and Lung Transplantation for Acute Cellular Rejection. Grading system has:
  * grade 0 (no acute rejection)
  * grade 1A (Focal, mild acute rejection)
  * grade 1B (Diffuse, mild acute rejection)
  * grade 2 (Focal, moderate acute rejection)
  * grade 3A (multifocal moderate rejection)
  * grade 3B (Diffuse, borderline severe acute rejection)
  * grade 4 (Severe acute rejection).
Time Frame: 6 months
Measure: Count of Units; unit: myocardial biopsies
Units Other Than Participants: myocardial biopsies
Arm/Group | Enteric-coated Mycophenolate Sodium (Myfortic)
Number analyzed (Participants) | 6
Number analyzed (myocardial biopsies) | 20
myocardial biopsies
  No rejection (Grade 0 or 1A) | 20
  Rejection (Grade 1B or higher) | 0
  Death due to rejection | 0

ADVERSE EVENTS:
Groups:
- Enteric-coated Mycophenolate Sodium (Myfortic): Enteric-coated Mycophenolate Sodium (Myfortic)
  1440mg/day (720mg by mouth, twice a day) of enteric-coated Mycophenolate Sodium (Myfortic) for 6 months
Arm/Group | Enteric-coated Mycophenolate Sodium (Myfortic)
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 8/11
Other Adverse Events (participants affected / at risk) | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enteric-coated Mycophenolate Sodium (Myfortic) (N=11)
Sepsis (Infections and infestations) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Heart re-transplant (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hypovolemia (Cardiac disorders) | 1 (1)
Steroid induced myopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
GI Bleeding (Gastrointestinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a small sample size study and 3 participants did not finish the 6 month visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No